CLINICAL TRIAL: NCT04274907
Title: A Phase 1b Study of Venetoclax in Combination With Pembrolizumab in Subjects With Previously Untreated NSCLC Whose Tumors Have High PD-L1 Expression
Brief Title: A Safety Study of Oral Venetoclax in Combination With Intravenous Pembrolizumab in Adult Participants With Previously Untreated Non-Small Cell Lung Cancer (NSCLC) With High Programmed Cell Death Ligand-1 (PD-L1) Expression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-700
Record Dates: First submitted 2020-02-17; First posted 2020-02-18 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer; Cancer
Keywords: Non Small Cell Lung Cancer (NSCLC); Cancer; Venetoclax; Pembrolizumab; PD-L1 Expression; ABT-199
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — venetoclax; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose Escalation Phase: Venetoclax + Pembrolizumab (Experimental): Participants will receive escalating doses of venetoclax in combination with pembrolizumab Dose A.
  Interventions: Drug: Venetoclax; Drug: Pembrolizumab
- Randomization Phase: Venetoclax + Pembrolizumab (Experimental): Participants will receive venetoclax at dose levels determined in the dose escalation phase in combination with pembrolizumab Dose A.
  Interventions: Drug: Venetoclax; Drug: Pembrolizumab
- Randomization Phase: Pembrolizumab Monotherapy (Active Comparator): Participants will receive pembrolizumab Dose A
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Venetoclax — Tablet: Oral
  Other Names: Venclexta; ABT-199
  Arms: Dose Escalation Phase: Venetoclax + Pembrolizumab; Randomization Phase: Venetoclax + Pembrolizumab
Drug: Pembrolizumab — Intravenous (IV) Infusion
  Other Names: Keytruda

SUMMARY:
Non-Small Cell Lung Cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. It is the most common form of lung cancer, accounting for around 85% of lung cancers. The purpose of this study is to evaluate the safety and efficacy (how well the study drug works against the disease) of venetoclax in combination with pembrolizumab in participants with NSCLC.

Venetoclax is a drug that kills cancer cells by blocking a protein (part of a cell) that allows cancer cells to stay alive. Pembrolizumab is approved drug for the treatment of NSCLC. It works with your immune system to help fight certain cancers. The study is split into two portions - dose escalation and randomization. Participants are assigned one of the three treatment groups to receive pembrolizumab alone or in combination with venetoclax. Each group receives a different treatment. Participants who are at least 18 years of age with a diagnosis of NSCLC will be enrolled. Around 100 participants will be enrolled in the study in approximately 44 sites across United States.

Participants will receive intravenous (IV) infusion of pembrolizumab alone or in combination with oral venetoclax tablets.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced or metastatic NSCLC with no known epidermal growth factor receptor (EGFR) sensitizing (activating) mutation or anaplastic lymphoma kinase (ALK) translocation.
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
* High PD-L1 tumor expression (tumor proportion score >= 50%) as determined by a Food and Drug Administration (FDA)-approved test.
* Willing to provide tissue biopsy sample prior to start of study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Received prior systemic treatment for their advanced or metastatic NSCLC. Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
* History of or ongoing interstitial lung disease or pneumonitis that required oral or intravenous (IV) steroids.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. If a participant has signs/symptoms suggestive of SARS-CoV-2 infection, they should undergo molecular (e.g., polymerase chain reaction [PCR]) testing to rule out SARS-CoV-2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to 28 Days
  DLTs are adverse events that are considered to have a reasonable possibility of relationship to the administration of venetoclax and pembrolizumab and cannot be attributed by the investigator to a clearly identifiable cause such as disease progression, concurrent illness or concomitant medication.
Change in the Sum of the Longest Diameter (SLD) | Up to 35 Cycles (Each Cycle is 21 Days)
  Change in the SLD is assessed by exposure-response modeling

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Venetoclax | Up to Cycle 1 (Each Cycle is 21 Days)
  Maximum plasma concentration (Cmax) of venetoclax
Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax | Up to Cycle 1 (Each Cycle is 21 Days)
  Time to maximum observed plasma concentration (Tmax) of venetoclax
Area Under the Plasma Concentration-Time Curve Over Time from 0 to 24 (AUC0-24) of Venetoclax in Plasma | Up to Cycle 1 (Each Cycle is 21 Days)
  Area Under the Plasma Concentration-time Curve (AUC) from 0-24 (AUC0-24)
Objective Response Rate (ORR) | Up to 35 Cycles (Each Cycle is 21 Days)
  ORR will be defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (39):
- United States (39):
  - Univ of Alabama at Birmingham /ID# 214180, Birmingham, Alabama
  - Arizona Oncology Associates, PC-HOPE (Rudasill) /ID# 216984, Tucson, Arizona
  - St Jude Hospital dba St Joseph /ID# 212360, Santa Rosa, California
  - Icri /Id# 217071, Whittier, California
  - AdventHealth Cancer Institute - Orlando /ID# 214444, Orlando, Florida
  - Georgia Regents University /ID# 217109, Augusta, Georgia
  - Rush University Medical Center /ID# 212448, Chicago, Illinois
  - University of Chicago DCAM /ID# 214319, Chicago, Illinois
  - Ingalls Memorial Hosp /ID# 214952, Harvey, Illinois
  - Fort Wayne Medical Oncology /ID# 214954, Fort Wayne, Indiana
  - Ashland-Bellefonte Cancer Ctr /ID# 218511, Ashland, Kentucky
  - University of Louisville /ID# 215195, Louisville, Kentucky
  - Central Maine Medical Center /ID# 216107, Lewiston, Maine
  - Maryland Oncology Hematology /ID# 214131, Columbia, Maryland
  - University of Massachusetts Ca /ID# 218744, Worcester, Massachusetts
  - Karmanos Cancer Institute /ID# 216986, Detroit, Michigan
  - Henry Ford Health System /ID# 216385, Detroit, Michigan
  - Univ of Mississippi Med Ctr /ID# 216429, Jackson, Mississippi
  - Washington University-School of Medicine /ID# 212355, St Louis, Missouri
  - Methodist Estabrook Cancer Center /ID# 216910, Omaha, Nebraska
  - University of Nebraska Medical Center /ID# 216754, Omaha, Nebraska
  - Hackensack Univ Med Ctr /ID# 216484, Hackensack, New Jersey
  - Atlantic Health System /ID# 217067, Morristown, New Jersey
  - Overlook Medical Center /ID# 219108, Summit, New Jersey
  - NYU Langone - Laura and Isaac Perlmutter Cancer Center /ID# 218077, New York, New York
  - Weill Cornell Medical Center /ID# 216911, New York, New York
  - University of Cincinnati Cancer Institute /ID# 216800, Cincinnati, Ohio
  - University Hospitals Cleveland /ID# 212241, Cleveland, Ohio
  - The Ohio State University - The James /ID# 212298, Columbus, Ohio
  - Providence Cancer Center Oncology and Hematology Care - Westside Portland /ID# 215497, Portland, Oregon
  - Allegheny General Hospital /ID# 214363, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Faris /ID# 217946, Greenville, South Carolina
  - Thompson Cancer Survival Ctr /ID# 217076, Knoxville, Tennessee
  - Houston Methodist Hospital - Scurlock Tower /ID# 215481, Houston, Texas
  - Utah Cancer Specialists /ID# 215496, Salt Lake City, Utah
  - Virginia Cancer Specialists /ID# 214328, Fairfax, Virginia
  - Massey Cancer Centre /ID# 212527, Richmond, Virginia
  - Multicare Institute for Research and Innovation /ID# 217913, Tacoma, Washington
  - Northwest Medical Specialties /ID# 218484, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/